CLINICAL TRIAL: NCT05307497
Title: An Exploration of Mother's Experiences of Antenatal Hand Expression of Colostrum, and the Effects Upon Breastfeeding Continuation and Maternal Emotional Health.
Brief Title: An Exploration of Antenatal Hand Expression.
Status: Completed | Type: Observational
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: 249857
Record Dates: First submitted 2022-03-10; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Feeding; Difficult, Newborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is an exploration of mother's experiences of antenatal hand expression of colostrum, and the effects upon breastfeeding continuation and maternal emotional health

DETAILED DESCRIPTION:
Second-line feeding strategies including hand expression and syringe feeding are used as an aid to breastfeeding, however little is known about their efficacy. This research explores the experiences of women who have used antenatal hand expression to identify how it affects maternal emotional health and breastfeeding continuation. UK women with recent experience of the practice were interviewed and the data analysed using thematic analysis. The results identified five themes in relation to these experiences including; The emotional distress of struggling with breastfeeding, Support as panacea but inconsistent, A crisis of confidence, Discord between knowledge, expectations and reality, and Syringe feeding as challenging but constructive. The study concludes that hand expression and syringe feeding supports women to establish breastfeeding, however, those struggling with breastfeeding need extra practical and emotional support to protect breastfeeding self-efficacy, emotional health and breastfeeding continuation. The findings highlight the importance of realistic, antenatal breastfeeding education to achieve this. Further research into second-line strategies and antenatal education programmes could contribute to the improvement of women's infant feeding experiences and improve UK breastfeeding rates.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18,
* Women with experience of antenatal hand expression within the last three months,
* Women with a good grasp of the English language.

Exclusion Criteria:

* Mothers of babies born before 37 weeks or with a medical issue (eg. tongue tie),
* Women with a mental health diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with experience of antenatal hand expression
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview | One hour
  Semi-structured interviews carried out with participants to collect qualitative data, analysed using thematic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT05307497/Prot_000.pdf